CLINICAL TRIAL: NCT05002036
Title: Evaluation of the Clinical Efficacy of Hyaluronic Acid and Gingko Biloba Eyedrops in the Management of Iatrogenic Dry Eye Disease Induced by Cataract Surgery
Brief Title: Management of Dry Eye Disease After Cataract Surgery With Topical Hyaluronic Acid and Gingko Biloba
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fogagnolo, Principal Investigator, Clinical Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCU-OS-003/2019
Record Dates: First submitted 2021-07-28; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA-GB (Active Comparator): eyedrop containing hyaluronic acid and gingko biloba (Trium eyedrops, Sooft srl)
  Interventions: Device: Trium eyedrops
- No treatment (No Intervention): no treatment for iatrogenic dry-eye

INTERVENTIONS:
Device: Trium eyedrops — given three times daily from day 1 after surgery to end of Week 4
  Arms: HA-GB

SUMMARY:
Cataract surgery is one of the main causes of Dry Eye Disease (DED). This paper aimed at evaluating the prevalence of iatrogenic DED on a population of patients without DED receiving cataract surgery, and the impact of an eyedrop containing hyaluronic acid and gingko biloba (HA-GB, Trium free eyedrops, Sooft srl, Italy).

In this phase-IV trial we enrolled 40 patients with no DED. Patients were seen at baseline, day 1, week 1 and week 4. At each visit patients received Ocular Surface Disease Index (OSDI) questionnaire, Anterior segment ophthalmoscopy with grading of conjunctival hyperemia, fluorescein tear break-up time (TBUT), grading of fluorescein corneal staining (epithelial damage); adherence and tolerability using a visual analogue scale were checked at week 1 and 4.

At day 0 patients underwent cataract surgery (2.4 mm temporal incision) and were randomized to standard postoperative care (control group) or standard postoperative care + HA-GB given three times a day for 4 weeks (HA-GB group).

ELIGIBILITY:
Inclusion criteria were:

* At least 18 years old Cataract requiring surgery
* TBUT of 7" or more in both eyes.

Exclusion criteria were:

* BUT of 6 seconds or less in one or both eyes
* Corneal staining of grade 2 or more using Oxford scale in one or both eyes
* Presence of corneal neuropathy (Cochet-Bonnet esthesiometry less than 50 mm) in one or both eyes
* Contact lens wear less than 30 days before surgery
* Neuropathic causes of dry eye (diabetes, long-standing contact lens wearing, previous ocular herpes infections)
* Autoimmune diseases
* Past or active ocular surface diseases (any corneal disease, cicatricial conjunctivitis, ocular surface burns, keratinization of the eyelid margin, Sjogren syndrome, corneal trauma)
* pregnant and lactating women pediatric patients or adolescents under 18 years
* ocular or general factors predisposing the patient to an increased risk for intraoperative complications, according to investigator's evaluation. These include (but are not limited to) pseudoexfoliation capsulae, complete cataract, iridodonesis, previous eye surgery, previous eye trauma, history of complicated cataract surgery in the fellow eye, benign prostatic hyperplasia under treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Tear Break-up time (TBUT), seconds | Changes occurring between Day 1 vs Week 1 and Week 4
  The time (seconds) from blinking from the first break of the tear film stained with fluorescein and evaluated at the slit lamp with blue cobalt filter and 10x magnification
Ocular Surface Disease Index (OSDI) | Changes occurring between Day 1 vs Week 1 and Week 4
  A score ranging from 0 to 100 calculated by means of a questionnaire

SECONDARY OUTCOMES:
Number of patients with TBUT of 5 sec or less | Changes occurring between Day 1 vs Week 1 and Week 4
Number of patients with corneal epithelial staining | Changes occurring between Day 1 vs Week 1 and Week 4
  Staining was evaluated at the slit lamp with fluorescein dying, blue cobalt filter and 10x magnification. Staining was graded according to the Oxford scale, ranging from 0 (no staining) to 4
Judgement of quality of study medications | Week 1, Week 4
  Patients were asked to judge the quality of study medications using a Visual analogue scale. The score was converted on a scale between 0 (very bad evaluation) and 100 (very high satisfaction)
Conjunctival hyperemia | Changes occurring between Day 1 vs Week 1 and Week 4
  Assessed using diffuse white illumination at the slit lamp with 10x magnification. Results were reported using Efron scale, ranging from 0 (normal) to 4 (severe)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fogagnolo P, Romano D, De Ruvo V, Sabella P, Rossetti L. Clinical Efficacy of an Eyedrop Containing Hyaluronic Acid and Ginkgo Biloba in the Management of Dry Eye Disease Induced by Cataract Surgery. J Ocul Pharmacol Ther. 2022 May;38(4):305-310. doi: 10.1089/jop.2021.0123. Epub 2022 Apr 18. PMID 35442771